CLINICAL TRIAL: NCT06086145
Title: Flavanol Intake in Davis (FID) Study: Biomarker-estimated Habitual (-)-Epicatechin and Flavanol Intake in Adults
Brief Title: Biomarker-estimated Flavanol Intake in Davis (FID)
Acronym: FID
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2052789
Record Dates: First submitted 2023-09-07; First posted 2023-10-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Diet; Adults
Keywords: Flavanols; Dietary flavanols; Phytonutrients; Bioactives; Observational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults in Davis and the greater Sacramento area of California: Adults in Davis and the greater Sacramento area of California
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Flavanols are compounds present in plants, including apples, berries, peaches, cocoa-derived products and certain beverages like tea. Following intake, they are absorbed and broken down into smaller compounds called 'metabolites'. Some of these metabolites are excreted in urine. In this study, we hope to collect urine and examine the metabolites to learn more about the types and amounts of flavanols that people are consuming as part of their usual diet.

DETAILED DESCRIPTION:
Flavanols, including the monomers (-)-epicatechin and (+)-catechin, and their related oligomeric derivatives, the procyanidins, are a group of plant-derived, dietary bioactives amply present in the diet. Supported by accumulating epidemiological studies and outcomes from the first large-scale randomized study with bioactives, the COcoa Supplement and Multivitamin Outcomes Study (COSMOS), the Academy of Nutrition and Dietetics released the first dietary recommendation for flavan-3-ols intake in the United States (US). This recommendation suggests the consumption of 400-600 mg/d of flavan-3-ols to mediate cardiometabolic beneficial effects, including the reduction of cardiovascular disease risk. While previous studies have aimed at assessing dietary intake of this group of bioactives, the tools used for these assessments were based on dietary questionnaires and food content databases. These tools are subjective and known to present significant limitations. Recently, our laboratory developed a series of nutritional biomarkers to objectively assess flavanol intake and thus, overcome limitations inherent to previous methods. These biomarkers are based on the quantification of a series of flavanol metabolites, including the 5-(3,4-dihydrophenyl)-γ-valerolactone metabolites (gVLM) and the structurally related (-)-epicatechin metabolites (SREMs). These biomarkers provide complementary information; as while gVLM provide information about the intake of flavanols in general, SREMs are specific biomarkers of (-)-epicatechin intake. In addition, gVLM are surrogate biomarkers, which means that this biomarker allows ranking volunteers from low to high flavanol consumers without providing information on absolute intake. On the other hand, SREMs proved to perform as a recovery biomarker when assessed in 24-hour urine, thus providing absolute amount of (-)-epicatechin consumed. While gVLM and SREM biomarkers have been used to assess the intake of flavanols and epicatechin in the United Kingdom, little is known about biomarker-estimated intake of flavanols in the US, and even less when considering the use of SREM as a recovery biomarker. Therefore, the characterization of flavanol and epicatechin intake in a US population will provide essential information to understand efforts to promote flavanol intake based on current dietary recommendations and thus increase access of the health benefit related to the consumption of these bioactives to the public in general.

ELIGIBILITY:
Inclusion criteria:

* 25 - 75 years old
* Male or female
* BMI 18.5 - 34.9 kg/m2
* Weight ≥ 110 pounds
* Computer, tablet or smart phone with cellular data/Wi-Fi to establish video call communication

Exclusion criteria:

* Adults unable to consent
* Prisoners
* Non-English speaking*
* BMI ≥ 35 kg/m2
* Indications of substance or alcohol abuse within the last 3 years
* Cancer of the GI tract, previous GI surgery (except appendectomy) or GI stoma
* History of difficult blood draws
* Diarrhea, defined as 3 or more loose or liquid stools/day, within the last 3 months or antibiotic intake within the last 3 months
* Currently participating in a clinical or dietary intervention study

  * Non-English speaking volunteers will be excluded for safety reasons, as we do not have staff that can adequately provide interpretation services that can explain and answer questions with regard to study procedures.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Free living adults in Davis and the greater Sacramento area of California.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Biomarker-estimated (-)-epicatechin and flavanol intake | 1 day
  Biomarker-estimated habitual (-)-epicatechin and flavanol intake assessed as the urinary concentration of SREM and gVLM in 24 hr urine.

SECONDARY OUTCOMES:
Subgroup analysis of biomarker-estimated (-)-epicatechin and flavanol intake by age, sex, anthropometric and clinical characteristics | 1 day
  Characterization of biomarker-estimated habitual (-)-epicatechin and flavanol intake (assessed as urinary concentrations of SREM and gVLM in 24 hr urine) by age, sex, anthropometric and clinical (health or disease status) characteristics.
Change of biomarker-estimated (-)-epicatechin and flavanol intake as a function of the intake of individual foods | 1 day
  Change of the biomarker-estimated habitual (-)-epicatechin and flavanol intake (assessed as the urinary concentration of SREM and gVLM in 24 hr urine) as a function of the intake of individual foods (assessed by the Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool).
Change of biomarker-estimated (-)-epicatechin and flavanol intake as a function of diet quality | 1 day
  Change of the biomarker-estimated habitual (-)-epicatechin and flavanol intake (assessed as the urinary concentration of SREM and gVLM in 24 hr urine) as a function of diet quality (assessed by food frequency questionnaire; Diet History Questionnaire III (DHQ III)).
Inter-day variation of biomarker-estimated (-)-epicatechin and flavanol intake | 1 day
  Inter-day variation of the biomarker-estimated habitual (-)-epicatechin and flavanol intake (assessed as the urinary concentration of SREM and gVLM in 24 hr urine) in a sub-cohort of volunteers.
Biomarker-estimated (-)-epicatechin and flavanol intake in spot urine | 1 day
  Biomarker-estimated habitual (-)-epicatechin and flavanol intake assessed as the urinary concentration of SREM and gVLM in spot urine.

OTHER OUTCOMES:
Blood pressure | 1 day
  Systolic and diastolic blood pressure will be measured as determined with SphygmoCor® XCEL.
Augmentation index | 1 day
  Augmentation index will be measured as determined with SphygmoCor® XCEL.
Lipid panel | 1 day
  Lipid panel will be assessed using validated methods by a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Francene M. Steinberg, PhD, RD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhagwat, S. and Haytowitz, D.B. (2015). USDA Database for the Proanthocyanidin Content of Selected Foods, Release 2 (2015). Nutrient Data Laboratory, Beltsville Human Nutrition Research Center, ARS, USDA. https://doi.org/10.15482/USDA.ADC/1324621.
- [Background] Bhagwat, S. and Haytowitz, D.B. (2016). USDA Database for the Flavonoid Content of Selected Foods. Release 3.2 (November 2015). Nutrient Data Laboratory, Beltsville Human Nutrition Research Center, ARS, USDA. https://doi.org/10.15482/USDA.ADC/1324465.
- [Background] Raman G, Avendano EE, Chen S, Wang J, Matson J, Gayer B, Novotny JA, Cassidy A. Dietary intakes of flavan-3-ols and cardiometabolic health: systematic review and meta-analysis of randomized trials and prospective cohort studies. Am J Clin Nutr. 2019 Nov 1;110(5):1067-1078. doi: 10.1093/ajcn/nqz178. PMID 31504087
- [Background] Sesso HD, Manson JE, Aragaki AK, Rist PM, Johnson LG, Friedenberg G, Copeland T, Clar A, Mora S, Moorthy MV, Sarkissian A, Carrick WR, Anderson GL; COSMOS Research Group. Effect of cocoa flavanol supplementation for the prevention of cardiovascular disease events: the COcoa Supplement and Multivitamin Outcomes Study (COSMOS) randomized clinical trial. Am J Clin Nutr. 2022 Jun 7;115(6):1490-1500. doi: 10.1093/ajcn/nqac055. PMID 35294962
- [Background] Crowe-White KM, Evans LW, Kuhnle GGC, Milenkovic D, Stote K, Wallace T, Handu D, Senkus KE. Flavan-3-ols and Cardiometabolic Health: First Ever Dietary Bioactive Guideline. Adv Nutr. 2022 Dec 22;13(6):2070-2083. doi: 10.1093/advances/nmac105. PMID 36190328
- [Background] Wang Y, Chung SJ, Song WO, Chun OK. Estimation of daily proanthocyanidin intake and major food sources in the U.S. diet. J Nutr. 2011 Mar;141(3):447-52. doi: 10.3945/jn.110.133900. Epub 2011 Jan 26. PMID 21270367
- [Background] Bai W, Wang C, Ren C. Intakes of total and individual flavonoids by US adults. Int J Food Sci Nutr. 2014 Feb;65(1):9-20. doi: 10.3109/09637486.2013.832170. Epub 2013 Sep 11. PMID 24020353
- [Background] Kuhnle GGC. Nutrition epidemiology of flavan-3-ols: The known unknowns. Mol Aspects Med. 2018 Jun;61:2-11. doi: 10.1016/j.mam.2017.10.003. Epub 2017 Nov 16. PMID 29146101
- [Background] Ottaviani JI, Fong R, Kimball J, Ensunsa JL, Britten A, Lucarelli D, Luben R, Grace PB, Mawson DH, Tym A, Wierzbicki A, Khaw KT, Schroeter H, Kuhnle GGC. Evaluation at scale of microbiome-derived metabolites as biomarker of flavan-3-ol intake in epidemiological studies. Sci Rep. 2018 Jun 29;8(1):9859. doi: 10.1038/s41598-018-28333-w. PMID 29959422
- [Background] Ottaviani JI, Fong R, Kimball J, Ensunsa JL, Gray N, Vogiatzoglou A, Britten A, Lucarelli D, Luben R, Grace PB, Mawson DH, Tym A, Wierzbicki A, Smith AD, Wareham NJ, Forouhi NG, Khaw KT, Schroeter H, Kuhnle GGC. Evaluation of (-)-epicatechin metabolites as recovery biomarker of dietary flavan-3-ol intake. Sci Rep. 2019 Sep 11;9(1):13108. doi: 10.1038/s41598-019-49702-z. PMID 31511603
- [Background] Ottaviani JI, Borges G, Momma TY, Spencer JP, Keen CL, Crozier A, Schroeter H. The metabolome of [2-(14)C](-)-epicatechin in humans: implications for the assessment of efficacy, safety, and mechanisms of action of polyphenolic bioactives. Sci Rep. 2016 Jul 1;6:29034. doi: 10.1038/srep29034. PMID 27363516
- [Background] Ottaviani JI, Britten A, Lucarelli D, Luben R, Mulligan AA, Lentjes MA, Fong R, Gray N, Grace PB, Mawson DH, Tym A, Wierzbicki A, Forouhi NG, Khaw KT, Schroeter H, Kuhnle GGC. Biomarker-estimated flavan-3-ol intake is associated with lower blood pressure in cross-sectional analysis in EPIC Norfolk. Sci Rep. 2020 Oct 21;10(1):17964. doi: 10.1038/s41598-020-74863-7. PMID 33087825

DOCUMENTS (1):
  • Informed Consent Form (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT06086145/ICF_000.pdf